CLINICAL TRIAL: NCT06567678
Title: The Effect of Colchicine on Platelet Function Profiles in Patients With Stable Coronary Artery Disease in Trinidad and Tobago. The Pilot ECLIPSE Study.
Brief Title: The Effect of Colchicine on Platelet Function Profiles in Patients With Stable Coronary Artery Disease
Acronym: ECLIPSE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of The West Indies (Other)
Responsible Party: Principal Investigator, Naveen Seecheran, Principal Investigator, The University of The West Indies
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CREC-SA2525/02/2024
Record Dates: First submitted 2024-08-20; First posted 2024-08-23 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Colchicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Colchicine 0.5mg po bd (Experimental): Patients with coronary disease taking Colchicine 0.5mg twice-daily orally for two weeks
  Interventions: Drug: Colchicine 0.5 MG oral tablet twice daily

INTERVENTIONS:
Drug: Colchicine 0.5 MG oral tablet twice daily — Blood samples will be collected from participants in 2 separate instances. Initially, a baseline VerifyNow P2Y12 PRU and Aspirin reaction unit test assay, followed by a subsequent repeat test 2-week after a 2-week, colchicine 0.5mg oral tablet twice-daily

SUMMARY:
The effects of colchicine on cardiovascular health in patients with stable coronary artery disease have been shown to be beneficial due to its anti-inflammatory properties. This present study aims to explore the effects of colchicine on platelet reactivity in patients with coronary artery disease on dual antiplatelet therapy.

DETAILED DESCRIPTION:
Recent landmark clinical trials on the use of colchicine in patients with chronic coronary artery disease has led to its implementation as an FDA approved drug for secondary prevention in patients with coronary artery disease. Colchicine exerts a range of anti inflammatory effects which plays a major role in reduction of atherosclerosis and prevention cardiovascular events. This current study aims to investigate the effect of colchicine on platelet reactivity in patients with stable coronary artery disease already on dual anticoagulants.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable coronary artery disease.
* Patients older than 18 years of age.
* Patients currently on dual anti platelets, aspirin and clopidogrel

Exclusion Criteria:

• Patients already on colchicine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2024-08-21 (Actual); Primary Completion 2024-10-20 (Actual); Study Completion 2024-11-04 (Actual)

PRIMARY OUTCOMES:
P2Y12 reaction units and Aspirin reaction units | two weeks
  P2Y12 and Aspirin reaction units pre and post colchicine 0.5mg twice daily oral dose.

CONTACTS AND LOCATIONS:
Overall Officials: Naveen Seecheran, Principal Investigator — The University of The west Indies, Saint Augustine, Trinidad and Tobago.
Locations (1):
- The University of The West Indies, Saint Augustine, Trinidad and Tobago

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available from the corresponding author on request.

REFERENCES:
- [Derived] Seecheran N, Grimaldos K, McCallum P, Ramcharan P, Kawall J, Katwaroo A, Grimaldos G, Seecheran V, Jagdeo CL, Rafeeq S, Seecheran R, Leyva Quert A, Ali N, Peram L, Motilal S, Ramtahal R, Bhagwandass N, Giddings S, Ramlackhansingh A, Sandy S. The Effect of Colchicine on Platelet Function Profiles in Patients with Stable Coronary Artery Disease: The ECLIPSE Pilot Study. Cardiol Ther. 2025 Mar;14(1):87-100. doi: 10.1007/s40119-024-00393-2. Epub 2025 Jan 18. PMID 39826082